CLINICAL TRIAL: NCT04699890
Title: Development of Specific Diagnostic Tools for Cardiac Insufficiency With Preserved Ejection Fraction
Acronym: MeDIAGSTOLE
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0466; 2020-A02216-33 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2020-09-21; First posted 2021-01-07 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
Keywords: Heart Failure (HF); progenitors cells; biomarkers; diastolic dysfunction
MeSH Terms: conditions — Heart Failure | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- preserved ejection fraction: Patients with a preserved ejection fraction (HF / FEp)
  Interventions: Other: Blood sampling, questionnaires and specific exams
- reduced ejection fraction: Patients with a reduced ejection fraction (HF / FEr)
  Interventions: Other: Blood sampling, questionnaires and specific exams
- without heart failure: Patient without heart failure
  Interventions: Other: Blood sampling, questionnaires and specific exams

INTERVENTIONS:
Other: Blood sampling, questionnaires and specific exams — Patients will have additionnal blood samples, answer to self-questionnaires and will performed an electrocardiogram and an echocardiography if not performed in routine care.

SUMMARY:
The MeDIAGSTOLE project aims to develop diagnostic tools for heart failure with preserved ejection fraction (IC / FEp), a pathology that is difficult to diagnose and to manage clinically in the absence of targeted treatment . The IC / FEp concerns the elderly population with comorbidities such as hypertension, obesity, anemia and atrial fibrillation. In the absence of specific biomarkers, clinical diagnosis is based on serum markers of heart failure with reduced ejection fraction (IC / FEr). The identification of new biomarkers, genetic and / or cellular, specific for IC / FEp would be an important innovation.

ELIGIBILITY:
Inclusion Criteria group 1 (ejection fraction ≥ 50%) :

* Age > or = 65,
* heart failure (NT-proBNP ≥ 450 pg/mL during hospitalization or follow-up)
* echocardiography showing an ejection fraction ≥ 50%,
* patients already hospitalized and followed in cardiology consultation,
* patients agreeing to sign informed consent,
* patient affiliated to french health care system.

Inclusion Criteria group 2 (ejection fraction < 50%) :

* Age > or = 65,
* heart failure (NT-proBNP ≥ 450 pg/mL during hospitalization or follow-up)
* echocardiography showing an ejection fraction < 50%,
* patients already hospitalized and followed in cardiology consultation,
* patients agreeing to sign informed consent,
* patient affiliated to french health care system.

Inclusion Criteria group 3 (without heart failure) :

* Age > or = 65,
* patients already hospitalized and followed in cardiology consultation for one of the following pathology : stable coronaropathy without heart failure, arterial hypertension without heart failure, auricular fibrilation without heart failure
* patients agreeing to sign informed consent,
* patient affiliated to french health care system.

Exclusion Criteria for all groups:

* Hemodynamic instability (cardiogenic shock),
* any condition leading to a prognosis of less than 7 days,
* Known hepatocellular insufficiency, or known hepatic cirrhosis
* ASAT / ALAT> 10N excluding cardiac cause
* Any conditions that may put the patient at risk or increase the risk of non-compliance with the protocol or lost to follow-up according to the opinion of the investigator
* Patient under legal protection, under guardianship or under curatorship
* Inability to give the subject informed information
* Pregnant or breastfeeding woman

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The inclusions will be done in the Cardiology department (Prof. F. Roubille) by the team of cardiologists trained in the study. Patients eligible for the study will be selected either from already hospitalized patients or from outside patients during the weekly consultation.
  In order to be representative of the population of interest (patients followed in cardiology consultation) and to limit inclusion bias, the inclusions will be exhaustive and consecutive. A collection of reasons for refusal will be made for the construction of the study flow chart.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
diagnostic power of a multi-marker approach (progenitor cells) | At 12 months
  to estimate the diagnostic power of a the multi-marker approach combining 5 circulating biomarkers (biochemical and cellular) in IC / FEp versus heart failure with reduced ejection fraction (IC / FEr) : first biomarker (cellular) : progenitor cells Value in µL.
diagnostic power of a multi-marker approach (monocytes) | At 12 months
  to estimate the diagnostic power of a the multi-marker approach combining 5 circulating biomarkers (biochemical and cellular) in IC / FEp versus heart failure with reduced ejection fraction (IC / FEr) : second biomarker (cellular) : monocytes Value in µL.
diagnostic power of a multi-marker approach (NT-proBNP) | At 12 months
  to estimate the diagnostic power of a the multi-marker approach combining 5 circulating biomarkers (biochemical and cellular) in IC / FEp versus heart failure with reduced ejection fraction (IC / FEr) : third biomarker (biochemical) : NT-proBNP Value in ng/L.
diagnostic power of a multi-marker approach (sST2) | At 12 months
  to estimate the diagnostic power of a the multi-marker approach combining 5 circulating biomarkers (biochemical and cellular) in IC / FEp versus heart failure with reduced ejection fraction (IC / FEr) : fourth biomarker (biochemical) : sST2 Value in ng/L.
diagnostic power of a multi-marker approach (PIIINP) | At 12 months
  to estimate the diagnostic power of a the multi-marker approach combining 5 circulating biomarkers (biochemical and cellular) in IC / FEp versus heart failure with reduced ejection fraction (IC / FEr) : fifth biomarker (biochemical) : PIIINP Value in ng/L.

SECONDARY OUTCOMES:
Variation in gene expression | At 12 months
  Carry out a molecular approach based on high throughput genetic sequencing. This will make it possible to determine the variations in gene expression : coding or not coding RNA.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Aguilhon, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU Montpellier, Montpellier, France